CLINICAL TRIAL: NCT07282808
Title: Focal or Radical Therapy: a Lesion-based Molecular Evaluation in Prostate Cancer
Acronym: FLAME-PC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Veracyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1018
Record Dates: First submitted 2025-11-20; First posted 2025-12-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: focal therapy; decipher; cryotherapy; irreversible electroporation; hifu; biomarker
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Focal Therapy, Low Transcriptomic Risk Cohort (Experimental): Low Transcriptomic Risk for recurrence after FT: Decipher GC Score <0.5; OR GC 0.5-0.85 and non PSC-LP subtype
  Interventions: Diagnostic Test: Molecular Evaluation for Risk of Recurrence after FT
- Radical Therapy, High Transcriptomic Risk Cohort (Experimental): High Transcriptomic Risk for recurrence after FT: Decipher GC 0.5-0.85 and PSC-LP subtype, or GC >0.85
  Interventions: Diagnostic Test: Molecular Evaluation for Risk of Recurrence after FT
- Focal Therapy, Unselected for Transcriptomic Risk of Recurrence (Historical) (No Intervention): From ProAMFocal (NCT06491056): Focal Therapy performed on all comers (no molecular evaluation) based on clinical criteria only (PSA ≤15 ng/ml, GG2-4, MRI lesion size ≤3ml for single and ≤1.5ml for two lesions, no gross EPE, determined to be completely ablatable).

INTERVENTIONS:
Diagnostic Test: Molecular Evaluation for Risk of Recurrence after FT — Low Risk - Decipher GC <0.5, OR GC 0.5-0.85 and non-PSC-LP subtype High Risk - Decipher GC 0.5-0.85 and PSC-LP subtype, OR GC>0.85
  Other Names: Decipher GC score; Transcriptomic Signature
  Arms: Focal Therapy, Low Transcriptomic Risk Cohort; Radical Therapy, High Transcriptomic Risk Cohort

SUMMARY:
Focal therapy (FT) is a new approach to treating localized prostate cancer. Instead of treating the entire prostate, it targets only the cancerous areas while preserving healthy tissue. This helps reduce side effects like urinary, sexual, and bowel problems.

In a prospective observational expansion of a phase II clinical trial (ProAMFocal), 80% of patients with small, localized prostate cancers treated with FT had no cancer recurrence at one year, and 70% at 3 years after treatment. The investigators studied the genetic makeup of each cancer, and found that certain genetic markers and cancer subtypes were better at predicting recurrence than standard clinical measures.

Based on this, the investigators are launching the FLAME-PC trial. In this study, all patients who qualify for FT will first undergo genetic profiling of their cancer. Patients with favorable profiles (low risk based on genetic markers) will receive FT, while those with high-risk profiles will be advised to undergo standard treatments like prostate removal or radiation.

The investigators current main goal is to test if genetic profiling can help us better select patients for FT. They believe that patients chosen using this method will have low recurrence rates (<10%) compared to those in their previous study (20-30%). FLAME-PC aims to show that personalized treatment based on genetic profiling can improve outcomes for prostate cancer patients, offering effective cancer control with fewer side effects.

DETAILED DESCRIPTION:
Prostate cancer is the leading male cancer in the developed world. However, most prostate cancers are indolent, with only a few being aggressive, or clinically significant (csPCa). Standard radical whole-prostate treatments are effective but result in significant urinary, sexual and bowel side effects. Focal Therapy (FT) is a novel strategy where just the area of csPCa is treated, leaving normal prostate tissue intact, reducing damage to surrounding structures, thus minimizing the morbidity of treatment. This strategy is feasible if the csPCa is early and limited to a lesion of small volume.

However, despite detailed imaging and histological sampling, a significant proportion of patients identified today for FT still experience cancer recurrence. The investigators have recorded a 19.1% csPCa recurrence rate 1 year, and 29.3% (cumulative) 3 years after FT in their NMRC-NIG-funded clinical trial (n=80) despite mapping out csPCa tumors in detail using high resolution (3 Tesla) multiparametric magnetic resonance imaging (mpMRI) and extensive biopsies. Interrogating these failures in their NMRC-TA project, they found that csPCa lesions that recurred had greater transcriptomic risk (genomic classifier [GC] score 0.60 vs 0.38, P=0.014), and were more likely to be of a luminal molecular subtype (prostate subtyping classifier luminal proliferative [PSC-LP]). The investigators hypothesize that patients with lesions that are high GC, and are PSC-LP should undergo standard radical therapy rather than FT.

FLAME-PC (Focal therapy or radical therapy: Lesion-based Molecular Evaluation in Prostate Cancer), aims to prospectively validate the stratification of csPCa patients to FT or radical therapy based on their genomic risk and molecular profiles. Patients deemed clinically suitable for FT based on imaging and biopsy, will be offered FT if they additionally have a GC score ≤0.5 or non-PSC-LP subtype, whereas those with a GC score >0.5 and PSC-LP subtype will be offered radical therapy instead.

The investigators Hypothesis is that patients stratified to receive FT in FLAME-PC based on their molecular profiles will have a better cancer outcome than a historical prospective cohort of patients undergoing FT based on clinical criteria only. If proven, this will be transformative as this will be the first evidence for the use of molecular profiling in prostate cancer treatment selection. Additionally, the investigators will gain further insights into the pre-FT molecular profiling (RNA analysis will be supported by and performed in collaboration with industry partner Veracyte, Inc.)

FLAME-PC is the first prospective trial to attempt to stratify early prostate cancer treatment between FT and radical therapy. This will provide the investigators with the opportunity to transform clinical paradigm of primary treatment selection in localized prostate cancer, lead to better patient cancer outcomes with FT, and reduce overall morbidity in patients suffering from prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Prostate Adenocarcinoma
* Grade Group 2-4
* MRI lesion size ≤3ml for single lesions ≤1.5ml for 2 lesions
* no gross EPE
* assessed to be completely ablatable with margin with focal therapy.

Exclusion Criteria:

* Grade Group 5 cancer
* gross EPE
* multifocal (>2) clinically significant prostate cancer
* unablatable location (very apical, basal tumors, or otherwise determined by procedurist).

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2048-09 (Estimated)

PRIMARY OUTCOMES:
1-year Post-Focal Therapy (FT) clinically significant cancer recurrence | 12 months after FT
  Recurrence of clinically significant prostate cancer infield or outfield at 12-month MRI and biopsy after focal therapy

SECONDARY OUTCOMES:
1 year Post-Focal Therapy Infield clinically significant cancer recurrence | 12 months after FT
  Recurrence of clinically significant cancer (≥GG2) within the treated area at 12 months MRI and biopsy
1 year Post-Focal Therapy Outfield clinically significant cancer recurrence | 12 months after FT
  Recurrence of clinically significant cancer (≥GG2) outside the treated area at 12 months MRI and biopsy
Failure-free survival | Over 20 years following enrolment
  salvage treatment, metastatic cancer, systemic treatment, or transition to watchful waiting.
Metastatic Cancer Free Survival | Over 20 years following enrolment
  Free from metastatic cancer on imaging, and/or PSA ≥50 ng/ml
Cancer-specific Survival | Over 20 years following enrolment
  Death from Prostate Cancer
Overall Survival | Over 20 years following enrolment
  Death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Kae Jack Tay, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD is available to bona fide investigators who wish to collaborate
Supporting Information: Study Protocol
Time Frame: 7 years from end of study
Access Criteria: via the principle investigator

REFERENCES:
- [Background] Tay KJ, Hong BH, Ong EHW, Tan KM, Pacho GC, Wong SJ, Tan YG, Law YM, Ngo NT, Tan PH, Yuen JSP, Ho HSS, Chen K, Peng J, Foo CWT, Sam XX, Tuan JKL, Kanesvaran R, Gupta RT, Rozen S, Polascik TJ, Liu Y, Proudfoot J, Davicioni E, Khor LY, Chua MLK. Transcriptomic predictors of prostate cancer recurrence following focal cryotherapy: a pooled analysis of phase II trial and prospective cohort data. J Natl Cancer Cent. 2025 May 29;5(5):515-523. doi: 10.1016/j.jncc.2025.04.002. eCollection 2025 Oct. PMID 41111925